CLINICAL TRIAL: NCT02926287
Title: Ambulatory Surgery for Urogenital Prolapse : a Pilot Study
Acronym: PCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-A01939-38
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Prolapse
Keywords: prolapse surgery; ambulatory surgery
MeSH Terms: conditions — Prolapse | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ambulatory surgery (Experimental): All the patients operated for pelvic organ prolapse during the study time will be recruited. All the patient eligible for an Ambulatory surgery will be discharged earlier.
  Interventions: Other: Ambulatory surgery

INTERVENTIONS:
Other: Ambulatory surgery — All patients who accepting participation to the study and operated for prolapse surgery, Patient eligible for Ambulatory surgery and return home on the same day if delivery criteria are satisfied ( Chung criteria+tsuccessful trial of void) Patient not eligible for Ambulatory surgery are included as control group
  Other Names: POQ

SUMMARY:
Main objective is evaluation of success rate of ambulatory surgery (AS) for pelvic organ prolapse (POP). All surgical approaches (laparoscopic, vaginal) are included in the study.

Secondary objectives are AS rate in the overall population and reasons for ineligibility or failure of ambulatory surgery.

This pilot study will evaluate the feasibility of AS for POP and identify pitfalls in AS.

A randomized control study will follow PCAP study.

DETAILED DESCRIPTION:
The prolapse surgery will be performed in 13% of women. Improved surgical and anesthetic techniques available makes this surgery to ambulatory care, while the latter is only slightly conducted in France.

Main objective is evaluation of success rate of ambulatory surgery (AS) for pelvic organ prolapse (POP). All surgical approaches (laparoscopic, vaginal) are included in the study.

Secondary objectives are AS rate in the overall population and reasons for ineligibility or failure of ambulatory surgery.

This pilot study will evaluate the feasibility of AS for POP and identify pitfalls in AS.

A randomized control study will follow PCAP study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Planned POP surgery
* Valid social insurance
* French spoken and written
* Informed consent signed
* No exclusion criteria

Exclusion Criteria:

* Refuse participation to study
* Pregnant or lactating woman
* Vulnerable people (Article L 1121-6 of the french code of public health)
* Major subject to legal protection or unable to consent (Article 1121-8 of the french code of public health )
* Participation in another protocol for less than 3 months
* Patient not presenting all the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Success rate of ambulatory surgery in patient operated for urogenital prolapse | After the 2 years of recruitment
  Success rate = (number of patients with period of hospitalization < 12 hours)/ (number of patients operated for prolapsus)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Courtieu, Principal Investigator — Clinique Beau Soleil

IPD SHARING:
Plan to Share IPD: No